CLINICAL TRIAL: NCT00063947
Title: A Phase I Study of OSI-774 in Combination With Gemcitabine and Radiation in Locally Advanced, Non-Operable Pancreatic Cancer
Brief Title: Erlotinib, Gemcitabine, and Radiation Therapy in Treating Patients With Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01439; 03-031; NCI-5441; CDR0000305855; MSKCC-03031; U01CA069856 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; Radiotherapy; Radiation

ARMS (1):
- Treatment (radiotherapy, gemcitabine, erlotinib hydrochloride) (Experimental): Chemoradiotherapy: Patients undergo radiotherapy 5 days a week for 5.5 weeks. Beginning on day 1 and continuing concurrently with radiotherapy, patients receive gemcitabine IV over 30 minutes twice weekly and oral erlotinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease proceed to maintenance therapy. Maintenance therapy: Beginning 4-7 weeks after the completion of chemoradiotherapy, patients receive maintenance chemotherapy comprising gemcitabine IV over 30 minutes on days 1 and 8 and oral erlotinib once daily. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of erlotinib when given together with gemcitabine and radiation therapy in treating patients with locally advanced unresectable pancreatic cancer. Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining erlotinib with gemcitabine may make the tumor cells more sensitive to radiation therapy and may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of erlotinib given concurrently with gemcitabine and radiotherapy in patients with locally advanced unresectable pancreatic cancer.

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. II. Determine, preliminarily, the antitumor efficacy of this regimen, in terms of response rate, in these patients.

III. Determine the time to tumor progression and overall survival of patients treated with this regimen.

OUTLINE: This is a non-randomized, open-label, dose-escalation study of erlotinib.

Chemoradiotherapy: Patients undergo radiotherapy 5 days a week for 5.5 weeks. Beginning on day 1 and continuing concurrently with radiotherapy, patients receive gemcitabine IV over 30 minutes twice weekly and oral erlotinib once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 10 patients receive treatment at that dose.

Patients are radiologically restaged 3-4 weeks after completion of radiotherapy. Patients with stable or responsive disease proceed to maintenance therapy. Patients whose imaging studies suggest a potential for curative resection are referred for a surgical evaluation before initiating maintenance therapy.

Maintenance therapy: Beginning 4-7 weeks after the completion of chemoradiotherapy, patients receive maintenance chemotherapy comprising gemcitabine IV over 30 minutes on days 1 and 8 and oral erlotinib once daily. Treatment repeats every 21 days for a total of 4 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 19-28 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced, unresectable disease, defined by all of the following:

    * Obvious encasement of the celiac, hepatic, or superior mesenteric artery
    * Encasement of the portal or superior mesenteric vein not amenable to surgical resection
    * Extrapancreatic extension with or without regional lymph node involvement
    * No evidence of distant metastatic disease by staging laparoscopy*
  * Locally recurrent disease after prior curative surgery allowed provided the following are true:

    * No prior chemotherapy or radiotherapy
    * No evidence of distant metastatic disease by staging laparoscopy*
* No islet cell pancreatic cancer or lymphoma or sarcoma of the pancreas
* Measurable or evaluable disease

  * Primary pancreatic tumor is considered evaluable and not measurable disease
  * Lymph node mass considered measurable disease
* No known brain metastases
* Performance status - ECOG 0-2
* More than 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* Creatinine clearance ≥ 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No abnormalities of the cornea based on history (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* No Crohn's disease or inflammatory bowel disease that would preclude undergoing external beam radiotherapy
* Able to tolerate oral medication
* No requirement for IV alimentation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* See Disease Characteristics
* No prior gemcitabine
* See Disease Characteristics
* See Disease Characteristics
* No prior epidermal growth factor receptor-targeting therapy
* No prior therapy for pancreatic cancer (except surgery)
* No concurrent commercial or other investigational agents or therapies intended to treat the malignancy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-05; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of erlotinib hydrochloride based on the incidence of dose-limiting toxicity (DLT) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 7.5 weeks

SECONDARY OUTCOMES:
Toxicity as assessed by CTCAE version 3.0 | 7.5 weeks
Response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 6 years
  Kaplan-Meier methods will be utilized to estimate the response duration.
Progression-free survival as assessed by RECIST | From the time of study enrollment until progression of disease is documented, assessed up to 6 years
  Kaplan-Meier methods will be utilized to estimate the progression-free survival.
Overall survival | From the time of study enrollment until the date of death, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States